CLINICAL TRIAL: NCT05630716
Title: Pilot Evaluation Using The Non-Invasive Cardiac Output Monitor (NICOM) for Goal-directed Fluid Resuscitation for Inpatients With Hypotension and/or Septic Shock
Brief Title: Non-Invasive Cardiac Output Monitor (NICOM) for Goal-directed Fluid Resuscitation for Inpatients With Hypotension and/or Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MEDICAL PROTOCOL
Record Dates: First submitted 2022-11-08; First posted 2022-11-30 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Hypotension; Septic Shock
MeSH Terms: conditions — Sepsis; Hypotension; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-Invasive Cardiac Output Monitor (NICOM) (Experimental): adult inpatients with sepsis associated with acute hypotension and/or evidence of septic shock
  Interventions: Device: NICOM

INTERVENTIONS:
Device: NICOM — non-invasive monitor capable of measuring cardiac output (CO) and cardiac index (CI), and stroke volume (SV) and stroke volume index (SVI) based on heart rate. The NICOM technology will be implemented by the Rapid Response Team providers (Advanced Practice Providers) and ICU nurses at FSH, most of whom are already trained and familiar with its use.

SUMMARY:
The Non-Invasive Cardiac Output Monitor (NICOM) is a non-invasive monitor capable of measuring cardiac output (CO) and cardiac index (CI), and stroke volume (SV) and stroke volume index (SVI) based on heart rate. Conceptually NICOM is a technology that utilizes a dynamic response characteristic in assessing the need for fluid administration, whereby SVI is measured before and after a fluid challenge with more fluid given only if SVI increases significantly with administered fluid. Dynamic response technologies are intended to replace older, "static" measures such as central venous pressure (CVP) and pulmonary capillary wedge pressures (PCWP) which are single point measurements utilized to assess the need to administer fluid.

The aim is to pilot and evaluate the effectiveness of using The Non-Invasive Cardiac Output Monitor (NICOM) technology for goal-directed fluid resuscitation in adult inpatients with sepsis associated acute hypotension and/or evidence of septic shock (Lactate >= 4.0).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients > 18 years of age
* inpatients for >/= 6 hours
* meeting criteria for sepsis as defined by hypotension related to sepsis (MAP < 65 or SBP < 90) or evidence of septic shock (Lactate ≥ 4.0).

Exclusion Criteria:

* Patients who die within 24 hours of hospital admission
* patients documented as "comfort cares" or enrolled in "general inpatient hospice" during the first 72 hours of hospitalization.
* opted out of having their medical information used in research, as noted in the EHR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | 18 months post-treatment
Hospital length of stay | 18 months post-treatment
ICU length of stay | 18 months post-treatment

SECONDARY OUTCOMES:
Hours of vasopressor use | 18 months post-treatment
change from baseline serum creatinine | 18 months post-treatment
Difference in positive fluid balance at 75 hours of ICU discharge | 75 hours post treatment ( ICU discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Dichter, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No